CLINICAL TRIAL: NCT04288050
Title: Evaluation of Glycemic Profiles in Diabetic Patients on Dialysis Under Insulin Balsal-bolus Protocol, Using Freestyle Libre. Observational Prospective Study Without Modification of Management.
Brief Title: Evaluation of Glycemic Profiles in Diabetic Patients on Dialysis Under Insulin Balsal-bolus Protocol, Using Freestyle Libre
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0586
Record Dates: First submitted 2019-12-04; First posted 2020-02-27 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Diabetic
Keywords: continuous glucose monitoring system; haemodialysis; peritoneal dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic subjects under dialysis: Diabetic subjects under dialysis

SUMMARY:
In France, chronic end-stage renal disease affects more than 11,000 new patients each year who will require dialysis or renal transplantation, of whom approximately 22.6% of new cases are related to diabetes. Among them, about 94% are managed by hemodialysis (HD), the others by peritoneal dialysis (PD). In addition, nearly 42% of dialysis patients have diabetes. There are issues related to glycemic control during dialysis and specific to each dialysis technique. Thus, hypoglycemic risk is the main risk observed during hemodialysis sessions, linked in particular to the use of a 1g/L glucose free dialysate, a decrease in renal neoglucogenesis and alterations in metabolic pathways. In addition, long-term glycemic control is difficult to assess in dialysis patients, because of the limitations of HbA1c witch is frequently underestimated.

This can be explained by 2 mechanisms:

* EPO treatment is associated with an increase in the proportion of young érythrocytes
* reduction in the lifetime of red blood cells reducing the duration of interaction between glucose and hemoglobin.

The results of studies conducted using continuous glucose measurements over a short period of time (48 hours to 5 days) suggest a benefit in using continuous glucose measurement to detect glycemic fluctuations during dialysis. To our knowledge, no studies have been conducted to evaluate longer-term glycemic control with this technology. In addition, the investigators now have the Freestyle, which allows us to record the continuous measurement of interstitial glucose over a longer period of time and is reimbursed for people on insulin basal-bolus protocol.

Thus, the investigators propose an observational study to evaluate glycemic control during dialysis sessions, but also to analyze the correlation between parameters measured with Freestyle and HbA1c measured routinely, according to the follow-up recommendations in diabetics.

DETAILED DESCRIPTION:
Data : patient data (clinical, biological and additional examinations) on a database registered at the University Hospital of Montpellier, on the secure server.

* Computerized medical records (DXcare) and consultation letters.
* Analysis of Freestyle data on a dedicated Freestyle View software, after downloading data on this software

Demographic characteristics: Age, gender Clinical history: Older diabetes, presence of diabetic retinopathy, diabetic maculopathy, microalbuminuria or proteinuria, older dialysis, type of dialysis, presence of ischemic heart disease, history of stroke, arteriopathy, gastroparesis, diabetic neuropathy, high blood pressure, hypercholesterolemia.

Treatments: diabetes, type of kidney replacement, other treatments

Biological assessment: Creatinemia, DFG, microalbuminuria, HbA1C, Hemoglobinemia, HDL, LDL, triglyceridemia, cholesterol, albuminuria/creatinuria ratio, proteinuria/creatinuria ratio

Patients will sign a non-opposition form.

ELIGIBILITY:
Inclusion criteria:

* Subjects over 18 years of age
* dialysis patients
* diabetics (any diabetes)
* any anti-diabetic treatment
* no objection form

Exclusion criteria:

* Objection of the subject
* Subject under guardianship or tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with dialysis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the time in range glycemic profile | 12 month
  Evaluate the time in range glycemic profile in diabetic patients undergoing dialysis

SECONDARY OUTCOMES:
Time above range of glycemic target | 6 month
  Time above range of glycemic target
Time below range of glycemic target | 6 month
  Time below range of glycemic target
Glucose management Indicator | 6 month
  Glucose management Indicator
Number of hypoglycemic events | 6 month
  Number of hypoglycemic events
mean number of scans on diabetic subjects in Dialysis. | 6 month
  mean number of scans on diabetic subjects in Dialysis.
Evaluate the Delta between measured HbA1c and GMI. | 6 month
  Evaluate the Delta between measured HbA1c and GMI.
Evaluate the correlation between average interstitial glucose measured at Freestyle and measured HbA1c. | 6 month
  Evaluate the correlation between average interstitial glucose measured at Freestyle and measured HbA1c.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC